CLINICAL TRIAL: NCT01810705
Title: A Multicenter, Open, Randomized, Controlled Phase IIb Trial Evaluating Efficacy and Tolerability of GRASPA (L-asparaginase Encapsulated in Red Blood Cells, Eryaspase) Plus Low-dose Cytarabine vs Low-dose Cytarabine Alone, in Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML) Elderly Patients, Unfit for Intensive Chemotherapy
Brief Title: GRASPA Treatment for Patients With Acute Myeloblastic Leukemia
Acronym: ENFORCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPA-AML2012-01
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Results first posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: myeloid; leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — eryaspase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GRASPA (Experimental): patients will receive one injection of GRASPA (100 IU/kg) after each course of low-dose cytarabine (see Arm "Control")
  Interventions: Drug: GRASPA
- Control (No Intervention): patients will receive successive courses of low intensive chemotherapy, as subcutaneous low-dose cytarabine 20mg twice daily for 10 days per course (from day 1 to day 10), each course occurring every 28 days, for a duration up to 24 months

INTERVENTIONS:
Drug: GRASPA — Patients receiving Intervention (experimental group) will be treated with one injection of graspa per cycle of treatment, each cycle during 28 days, for a duration up to 24 cycles maximum
  Other Names: L-asparaginase encapsulated in red blood cells
  Arms: GRASPA

SUMMARY:
The protocol aims at adding GRASPA (L-asparaginase encapsulated in red blood cells, eryaspase) to standard chemotherapy (low-dose cytarabine) to treat patients older than 65 years diagnosed with AML and unfit for intensive chemotherapy.

DETAILED DESCRIPTION:
L-asparaginase (ASNase) holds a key role in chemotherapy for Acute Lymphoblastic Leukemia (ALL) in children and young adults. In elderly patients, its efficacy is counterbalanced by its toxicity, which impairs its use. However, a study conducted with GRASPA (L-asparaginase encapsulated in red blood cells, eryaspase) in elderly ALL (study reference "GRASPALL-GRAAL SA2 2008") showed that efficacy/safety profile was positive, paving the way for introducing ASNase benefit into chemotherapy for elderly patients.

In adults, Capizzi (1988) reported a significant benefit of ASNase associated with high-dose cytarabine treatment (HiDAC) in Acute Myeloid Leukemia (AML). Indeed, there was an overall statistically superior complete remission rate for HiDAC/ASNase (40%) vs HiDAC (24%) and an overall survival benefit for patients treated with HiDAC/ASNase (19.6 weeks vs 15.9 weeks).

Another study in elderly patients also displayed positive results for ASNase treatment (Petti, 1989), as well as recent single case reports that point out the potential benefit of ASNase in different AML or mixed lineage leukemia (Horikoshi, 2009; Rubnitz, 2009).

Our preclinical results also showed that an AML cell line and blast cells from the bone marrow of AML patients were sensitive to ASNase in vitro.

However, up to now, the toxicity of ASNase for elderly had prevented its use in this population that represents the majority of AML patients.

Considering the promising results of ASNase for AML treatment and the better safety profile offered by GRASPA (L-aspariginase encapsulated in red blood cells, erysapase), a multicenter, randomized, controlled IIb trial is open for recruitment. Efficacy and tolerability of GRASPA plus low-dose cytarabine will be evaluated versus low-dose cytarabine alone in treatment of AML patients over 65 year-old, unfit for intensive chemotherapy.

One hundred and twenty-three patients (65-85 year-old) newly diagnosed for AML are planned for inclusion in the study.

A 2:1 randomization will be respected (82 patients treated with GRASPA® plus low-dose cytarabine and 41 patients treated with low-dose cytarabine alone). Each patient will be followed for 24 months.

ELIGIBILITY:
Inclusion criteria:

* Patient > 65 years old and < 85 years old
* Newly diagnosed Acute Myeloid Leukemia (AML) or post myelodysplastic syndrome diagnosed within 6 months prior to study enrollment
* Unfit for intensive chemotherapy (at risk to suffer treatment related pejorative toxicities /early death) due to the presence of one or more of the following criteria: Dependence in activities of daily living owing to the presence of comorbidities other than those resulting from the deterioration caused by the neoplastic disease. Presence in the patient's medical history of three or more of the following comorbidities, even if they are under control with proper treatment: Congestive heart failure, other chronic cardiovascular diseases, chronic obstructive pulmonary disease, cerebrovascular disease, peripheral neuropathy, chronic kidney failure, hypertension, diabetes mellitus, systemic vasculitis, severe arthritis
* Presence of geriatric syndromes such as fecal or urinary incontinence, spontaneous bone fractures, mild and moderate dementia, or patients who fall repeatedly, or, patient unwilling to receive intensive chemotherapy
* Eligible to receive low-dose cytarabine treatment
* ECOG performance status ≤ 2
* Female patients of childbearing potential and males must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment and for 6 months after the last dose of Cytarabine or 3 months after last dose of GRASPA (whichever is the longest).
* Negative serum pregnancy test at study entry for female subjects of childbearing potential
* Subscription to social security insurance (if applicable, in accordance with local regulations)
* Ability to understand, and willingness to sign, a written informed consent document and to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion criteria:

* Patients with M3 AML of FAB classification (APL, acute promyelocytic leukemia)
* Patients with AML involving chromosome 16 abnormalities or translocation (8:21) (CBF-AML)
* Patient with secondary AML subsequent to prior malignant blood disorder such as: Myelodysplastic syndrome diagnosed more than 6 months before study entry or Myeloproliferative syndrome
* Prior therapy to AML (standard therapy or investigational agents)
* Inadequate organ function : Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis, Serum creatinine concentration > 2 x ULN (Upper Limit of Normal), AST or ALT levels > 3.5xULN or 5xULN if related to AML, Total bilirubin > 2 x ULN, INR > 1.5, unless patient under chronic treatment with anticoagulants (in this case, INR should be within expected ranges for the specific condition), Insulin-dependent or uncontrolled diabetes mellitus
* Concurrent malignancies other than AML requiring chemotherapy
* Severe active infection, HIV seropositivity, or known active type B or C viral hepatitis
* Known or suspected hypersensitivity or intolerance to mannitol
* Breastfeeding or lactating women

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: X Thomas, Doctor, Principal Investigator
Locations (21):
- France (21):
  - Hôpital l'Archet 1, Nice, Alpes Maritimes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Centre hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Institut Paoli Calmettes, Marseille, Bouche Du Rhone
  - Hôpital JEAN MINJOZ, Besançon, Doubs
  - Hopital Morvan, Brest, Finistere
  - Hôpital Haut-Lévèque, Pessac, Gironde
  - CHRU de Nîmes, Nîmes, Guard
  - Hopital de Hautepierre, Strasbourg, Haut Rhin
  - Hopital De Purpan CHU Toulouse, Toulouse, Haute Garonne
  - Hopital Région d'Annecy, Pringy, Haute Savoie
  - Hôpital Saint Eloi, Montpellier, Hérault
  - Hôtel Dieu - CHU de NANTES, Nantes, Loire Atlantique
  - Chu D'Angers, Angers, Maine Et Loire
  - Hopital de Brabois, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Hôpital Claude-Huriez, Lille, Nord
  - Institut de Cancérologie de la Loire, Saint-priest-en-jarez, Pays de la Loire Region
  - CHU Estaing, Clermont-Ferrand, Puy De Dome
  - hopital de Perpignan, Perpignan, Pyrénées Orientales
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - Groupe Hospitalier Sud, Amiens, Somme

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GRASPA | Control
Started | 83 | 40
Completed | 10 | 5
Not Completed | 73 | 35

BASELINE CHARACTERISTICS:
Groups:
- GRASPA: In the experimental group, the patients will receive one administration of GRASPA (100 IU/kg) at Day 11 in combination with subcutaneous low-dose cytarabine as 40 mg daily (either one single dose of 40 mg or 20 mg twice daily according to local practice) for 10 consecutive days, every 28 days, for duration up to 24 months
- Control: In the control arm, patients will be treated with subcutaneous low-dose cytarabine as 40 mg daily (either one single dose of 40 mg or 20 mg twice daily according to local practice) for 10 consecutive days, every 28 days, for duration up to 24 months. Each period of 28 days constitute a cycle of chemotherapy.
- Total: Total of all reporting groups
Arm/Group | GRASPA | Control | Total
Number analyzed (Participants) | 83 | 40 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 83 | 40 | 123
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 16 | 53
  Male | 46 | 24 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: OS is defined as the time elapsed between randomization and death from any cause.
Time Frame: Each patient will be followed for a duration of 24 months.
Population: OS was to be assessed by measuring time elapsed between randomisation and death for any cause. Any patient not known to have died at the time of analysis is censored based on the last recorded date on which the patient was known to be alive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GRASPA | Control
Number analyzed (Participants) | 83 | 40
months | 4.8 [3.1 to 7.0] | 6.4 [3.6 to 10.7]

2. Secondary Outcome: Response to Treatment
Description: Percentage of patients with Complete remission (CR), Complete remission with incomplete recovery (neutrophil or platelet regeneration, CRi), Partial remission (PR)
Time Frame: Each patient will be followed for a duration of 24 months.
Reporting Status: Not Posted

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time elapsed between randomization and resistant disease or relapse or death from any cause
Time Frame: Each patient will be followed for a duration of 24 months.
Reporting Status: Not Posted

4. Secondary Outcome: Patient Quality of Life
Description: Collecting survey about patients quality of life
Time Frame: Each patient will be followed for a duration of 24 months.
Reporting Status: Not Posted

5. Secondary Outcome: Safety of GRASPA Adverse Events and Serious Adverse Events
Description: Number of incidences, type, severity and causality of adverse events / serious adverse events
Time Frame: Each patient will be followed for a duration of 24 months.
Reporting Status: Not Posted

6. Secondary Outcome: Relapse Free Survival
Description: Defined only for patients who achieve CR or CRi as the time elapsed between date of CR/CRi and date of disease relapse or death from any cause
Time Frame: Each patient will be followed for a duration of 24 months.
Reporting Status: Not Posted

7. Secondary Outcome: Number of Hospitalizations
Description: Hospitalizations (except schedule protocol visit during the study)
Time Frame: Each patient will be followed for a duration of 24 months.
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Patients Who Need Transfusions
Description: Number of transfusions per patient (red blood cells and or platelets)
Time Frame: Until patient stops treatment (expected average of 8 months)
Reporting Status: Not Posted

9. Secondary Outcome: Pharmacodynamic and Pharmacokinetic Parameters of GRASPA
Description: Plasma concentrations of asparagine, aspartate, glutamine, glutamate, whole blood L- asparaginase activity
Time Frame: Until patient stops treatment (expected average of 8 months)
Reporting Status: Not Posted

10. Secondary Outcome: Immunogenicity
Description: Titer of anti L-asparaginase antibodies
Time Frame: Until patient stops treatment (expected average of 8 months)
Reporting Status: Not Posted

11. Secondary Outcome: Asparagine Synthetase (Optional)
Description: Asparagine synthetase and in vitro sensitivity to aspariginase on the harvested bone marrow cells
Time Frame: Until patient stops treatment (expected average of 8 months)
Reporting Status: Not Posted

12. Secondary Outcome: Biomarker Cytogenetic Testing (Optional)
Description: Defined as cytogenetic biomarker testing
Time Frame: Until patient stops treatment (expected average of 8 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signature of the informed consent from first patient and until 4 months after last GRASPA/ low-dose cytarabine administration of last patient i.e. up to 28 months for the longuest study drug exposure and on a total of 46 months of AE collection period throughout the study.
Groups:
- GRASPA: Patients having received at least one injection of GRASPA (100 IU/kg) i.e. 81 in GRASPA arm
- Control: Patients having received at least one dose of study treatment i.e. 39 in control arm
Arm/Group | GRASPA | Control
All-Cause Mortality (participants affected / at risk) | 70/81 | 34/39
Serious Adverse Events (participants affected / at risk) | 74/81 | 32/39
Other Adverse Events (participants affected / at risk) | 80/81 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRASPA (N=81) | Control (N=39)
Hypersensitivity (Immune system disorders) | 6 (6) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 8 (8) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 3 (5)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 1 (1)
Hemorrhagic Events (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 5 (7) | 1 (1)
General physical health deterioration (General disorders) | 10 (12) | 2 (2)
Pyrexia (General disorders) | 7 (7) | 2 (2)
Sepsis (Infections and infestations) | 12 (13) | 6 (6)
Septic shock (Infections and infestations) | 7 (7) | 6 (6)
Bronchopulmonary aspergillosis (Infections and infestations) | 4 (5) | 2 (2)
Lung infection (Infections and infestations) | 1 (2) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRASPA (N=81) | Control (N=39)
Epistaxis (Vascular disorders) | 10 (12) | 6 (6)
Hypertension (Vascular disorders) | 10 (12) | 4 (5)
Purpura (Vascular disorders) | 5 (5) | 2 (2)
Haematoma (Vascular disorders) | 4 (4) | 2 (2)
Petechiae (Vascular disorders) | 3 (3) | 2 (2)
Alloimmunisation (Immune system disorders) | 16 (16) | 1 (1)
Alloimmunisation (Immune system disorders) | 5 (5) | 2 (2)
Hypersensitivity (Immune system disorders) | 8 (14) | 0 (0)
asthenia (General disorders) | 28 (34) | 18 (20)
asthenia (General disorders) | 13 (17) | 9 (10)
Pain (General disorders) | 8 (8) | 2 (2)
Injection site haematoma (General disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 26 (50) | 13 (27)
General physical health deterioration (General disorders) | 4 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 11 (12) | 4 (4)
Depression (Psychiatric disorders) | 5 (5) | 3 (3)
Confusional state (Psychiatric disorders) | 4 (5) | 0 (0)
fall (Injury, poisoning and procedural complications) | 10 (12) | 3 (3)
Transfusion reaction (Injury, poisoning and procedural complications) | 7 (8) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Food poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood albumin decreased (Investigations) | 24 (29) | 6 (8)
Pancreatic enzymes abnormal (Investigations) | 20 (31) | 5 (5)
Transaminases increased (Investigations) | 15 (40) | 6 (10)
Antithrombin III decreased (Investigations) | 17 (22) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 15 (18) | 5 (5)
Weight decreased (Investigations) | 8 (9) | 7 (7)
Blood Creatinine increased (Investigations) | 12 (15) | 3 (3)
Blood chloride increased (Investigations) | 11 (15) | 2 (3)
Blood urea increased (Investigations) | 9 (9) | 4 (6)
Blood lactate dehydrogenase increased (Investigations) | 7 (8) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 3 (3)
Blood chloride decreased (Investigations) | 5 (6) | 3 (3)
Prothrombin time ratio decreased (Investigations) | 8 (10) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 6 (7) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac failure (Cardiac disorders) | 4 (4) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 59 (149) | 32 (84)
Leukopenia (Blood and lymphatic system disorders) | 41 (87) | 19 (31)
Neutropenia (Blood and lymphatic system disorders) | 35 (98) | 18 (34)
Lymphopenia (Blood and lymphatic system disorders) | 8 (9) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 8 (8) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 62 (170) | 34 (74)
Hemorrhagic Events (Blood and lymphatic system disorders) | 21 (23) | 9 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 12 (13) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 24 (57) | 15 (21)
Diarrhoea (Gastrointestinal disorders) | 24 (32) | 10 (12)
Constipation (Gastrointestinal disorders) | 18 (22) | 10 (11)
Vomiting (Gastrointestinal disorders) | 14 (27) | 5 (14)
Stomatitis (Gastrointestinal disorders) | 7 (7) | 3 (4)
Aphthous ulcer (Gastrointestinal disorders) | 9 (11) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (4)
Haemorrhoids (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 15 (25) | 5 (5)
Hepatocellular injury (Hepatobiliary disorders) | 5 (5) | 1 (2)
Renal failure (Renal and urinary disorders) | 12 (13) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 8 (10) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (19) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (10) | 3 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 (9) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT01810705/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT01810705/SAP_001.pdf